CLINICAL TRIAL: NCT03282942
Title: Effects of Aerobic or Strength Training on Cardiovascular, Endothelial Response, and Blood Flow in Hypertensive Middle Ages Individuals: a Randomized Controlled Clinical Trial.
Brief Title: Cardiovascular Effects of Aerobic and Strength Training in Hypertensive Middle-aged Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alvaro Reischak-Oliveira, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 69373217.3.0000.5347
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Arterial Hypertension
Keywords: hypertension; Aerobic training; Strength training
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training protocols (Experimental): Participants will be randomized in one of TWO groups: aerobic training group (AT) or strength training group (ST). Each training protocol will last 12 weeks, being the initial two weeks designed to participants' gradual adaptations to respective training protocol, with sessions performed three times per week in non-consecutive days.
  Interventions: Other: Strength training group; Other: Aerobic Training Group
- Control Group (No Intervention): The individuals who will be part of the control group will be instructed to follow their daily activities, avoiding any systematic exercise program and return to the end of the 12 weeks for reevaluation.

INTERVENTIONS:
Other: Strength training group — Individuals in the strength training group will perform exercises based on exercises with free weights and equipment, for upper and lower limbs with a weekly frequency of three times for twelve weeks. The periodization will start with 2 sets, 15 - 20 repetitions, passive rest of 120 seconds, exercises performed alternating by segments and the intensity of 50% of maximum repetition. After twelve weeks the periodization will be finished with 3 sets, 8-12 repetitions, passive rest of 120 seconds, exercises performed alternated by segments and the intensity of 70% of maximum repetition.
  The following exercises will compose the strength training protocol:
  * Squatting
  * Leg press
  * Knee Extension
  * Knee Flexion
  * Supine Challenge
  * High Pull
  * Elbow flexion
  * Extension of elbows
  * Development
  * Abdominal
  Arms: Exercise training protocols
Other: Aerobic Training Group — Individuals in the aerobic training group will perform aerobic treadmill exercise three times a week for twelve weeks. The training prescription will be performed through the percentage of maximum oxygen consumption with intensity in 60% to 80% with an average duration of 50 minutes of continuous exercise.
  Arms: Exercise training protocols

SUMMARY:
Systemic arterial hypertension (SAH) is characterized by elevated and sustained blood pressure levels, related to several risk factors. Modifying lifestyle to combat risk factors associated with cardiovascular disease is critical, as such factors are related alteration of endothelial vasodilator response leading to progressive loss of its protective function. However, endothelial dysfunction related to hypertension is not only related to the decrease in the bioavailability of endothelium relaxants, but also to the time of presence of hypertension, increased production of vessel contraction factors and oxidative stress related to the disease. In this way, physical training presents as a non-drug strategy capable of directly and indirectly influencing the pathophysiology of hypertension. In this way the objective of the present work will be to evaluate the acute and chronic effect of aerobic exercise and strength on blood pressure, blood markers of vasodilation and vascular endothelial vasoconstriction, as well as the repercussion on flow-mediated dilatation and oxidative stress markers, In middle-aged hypertensive individuals before and after 12 weeks of training. Study hypothesis: The expected results of the research are that the endothelial response of biochemical markers of vasodilation and vasoconstriction will change positively after aerobic and strength training and the responses will be similar when compared between groups. There will be an improvement in the antioxidant capacity in both groups and the magnitude of the hypotensive effect will be greater in the aerobic group when compared to control and strength.

ELIGIBILITY:
Inclusion Criteria:

Study inclusion criteria consisted of the following: 1) Individuals should use antihypertensive medication; 2) 30-59 years of age.

Exclusion Criteria:

The following aspects were regarded as exclusion criteria: 1) body mass index (BMI) up to 40 kg/m2; 2) regular engagement in any type of physical exercise training in the past 6 months prior to inclusion in the study; 3) symptomatic peripheral arterial occlusive disease; 4) aortic insufficiency or stenosis more than stage I; 5) hypertrophic obstructive cardiomyopathy; 6) congestive heart failure (>NYHA II); 7) uncontrolled cardiac arrhythmia with hemodynamic relevance; 7) change of antihypertensive medication in the past 4 weeks prior to inclusion in the study; 8) indication of unstable coronary artery disease. 9) use of tobacco products.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | End of 12-week exercise period
  24-h Ambulatory blood pressure
Endothelial Function | End of 12-week exercise period
  Flow mediated dilation to reactive hyperemia
Endothelium derived factors | End of 12-week exercise period
  The plasma levels of NOx and ET-1 will be determined by enzyme-linked immunosorbent assay
Inflammatory Profile | End of 12-week exercise period
  The inflammatory profile was accessed trough the cytokines and chemokines levels

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Reischak-Oliveira, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Ramis TR, Boeno FP, Leal-Menezes R, Munhoz SV, Farinha JB, Ribeiro JL, Reischak-Oliveira A. Effects of exercise modalities on decreased blood pressure in patients with hypertension. Front Physiol. 2022 Oct 14;13:993258. doi: 10.3389/fphys.2022.993258. eCollection 2022. PMID 36311227